CLINICAL TRIAL: NCT07150611
Title: A Multi-Perspective Interpretative Phenomenological Analysis of Patient and Bed Partner Experiences With CPAP Therapy Adaptation in Obstructive Sleep Apnoea
Brief Title: OSA Patients' and Bed-Partners' Illness Perceptions in CPAP Therapy Adaptation Process
Acronym: CPAP-IPA
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Eleonora Volpato, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: 04_26/04/2023
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: OSA - Obstructive Sleep Apnea
Keywords: Illness Perceptions; Bed Partners; OSA; CPAP therapy; CPAP adaptation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- T0-OSA Patients: OSA patients who are to be started on CPAP therapy but have not yet begun the adaptation process.
- T1-OSA Patients: OSA patients in their first year of CPAP adaptation.
- T2-OSA Patients: Patients who have been adapted to CPAP for over a year.
- T0-BedPartner: Bed partners of OSA patients who have to be adapted to CPAP therapy
- T1-BedPartner: Bedpartners of OSA patients in their first year of CPAP adaptation.
- T2-Bedpartner: bedpartners of patients who have been adapted to CPAP for over a year.

SUMMARY:
This study explores how psychological and relationship factors influence the success of CPAP therapy in people with Obstructive Sleep Apnea (OSA) and their partners. CPAP therapy is a common treatment for OSA, yet many patients struggle to keep using it consistently. Our research aims to identify what helps or hinders patients and their partners in adhering to CPAP therapy, including their illness perceptions, how they cope with treatment and how their relationship dynamics affect their experience. By understanding these factors, we hope to provide valuable insights to better support both patients and their bed partners, leading to improved treatment adherence and quality of life for couples managing OSA.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common condition that disrupts sleep due to repeated interruptions in breathing, which can lead to daytime fatigue, mood issues, and health risks like heart disease. Continuous Positive Airway Pressure (CPAP) therapy is the primary treatment, helping keep airways open during sleep and improving overall health. However, despite its benefits, many people find CPAP difficult to use consistently. Patients may feel uncomfortable or self-conscious about wearing the device, particularly around their partners, which can impact their relationships and adherence to treatment.

This study takes a unique approach by examining how OSA and CPAP therapy impact not only patients but also their "bed partners"-typically a spouse or close companion who shares their sleeping environment. Bed partners often play a supportive role, helping the patient manage OSA and adjust to CPAP therapy. Yet, little research has focused on how the partner's involvement, perceptions, and reactions influence the patient's experience and adherence to treatment.

Using the Interpretative Phenomenological Analysis (IPA) methodology with a Multi-Perspective approach, this study enables a dual view on the experiences of both patients and bed partners, offering an in-depth look at their shared journey with CPAP. Participants are recruited from the Sleep Medicine Clinic at Don Gnocchi in Milan and divided into three subgroups based on their stage in the CPAP adaptation process: T0, pre-adaptation; T1, within the first year of adaptation; and T2, following the first year of adaptation. This division allows for a nuanced understanding of how attitudes and experiences with CPAP may evolve over time.

Our study examines the psychological and relational aspects that affect CPAP adherence, seeking to uncover both the challenges and supports involved. Using the Common Sense Model of Illness Representation as a theoretical framework, we explore how the patient's and partner's understanding of OSA and CPAP can shape their responses and behavior. This model suggests that how people perceive an illness can strongly affect their actions, including their coping strategies. By studying both the patient's and partner's views, we aim to identify areas of potential miscommunication or stress that may hinder adherence and to find ways for healthcare providers to offer targeted support.

By focusing on the relationship between patients and bed partners, this study seeks to enhance our understanding of the social and emotional dynamics around CPAP therapy, which could lead to improved patient adherence and well-being.

ELIGIBILITY:
For patients:

Inclusion Criteria:

* Adult partcipants with mild (Apnea/Hypopnea Index, AHI between 5 and 15), moderate (AHI between 15 and 30), or severe (AHI greater than 30) OSA (Young et al., 2009), as certified by a pulmonologist at the recruitment centre, with a stable bed partner;
* Participants with OSA awaiting CPAP therapy initiation, or those who are either adherent or non-adherent within the first year of CPAP use or who have been using CPAP for over a year;
* Participants who provided informed consent to participate in the study;
* Participants who are proficient in the Italian language.

Exclusion Criteria:

* Participants who did not provide informed consent to participate;
* Participants who do not speak Italian;
* Participants who have not been diagnosed with OSA and for whom CPAP therapy is not deemed necessary or who are not currently undergoing CPAP therapy;
* Participants with OSA without a stable bed partner;
* Participants with significant psychiatric comorbidities or with other significant organic pathologies where OSA is not the primary health concern, according to medical records;

For bedpartners

Inclusion criteria:

* Bed partners in a stable relationship with an OSA patient for whom CPAP therapy adaptation has been deemed necessary or who are already adapted to CPAP therapy;
* Bed partners who have provided informed consent to participate;
* Bed partners who are proficient in the Italian language.

Exclusion criteria:

* Bed partners who did not provide informed consent;
* Bed partners who do not speak Italian;
* Bed partners without a stable relationship with an OSA patient for whom CPAP therapy adaptation has been deemed necessary or who are already adapted to CPAP therapy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive Sleep Apnea (OSA) patients and their bed partners at 3 different step of OSA management. The subgroups included:
  * (1) OSA patients and bed partners before starting CPAP therapy (T0)
  * (2) OSA patients and bed partners within the first year of CPAP use (T1)
  * (3) OSA patients and bed partners beyond one year of CPAP use (T2).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Experience of CPAP usage and adaptation and lived OSA condition | From enrollment to the end of the interviews one week later
  A multi-perspective (patients and bed partners) interpretative phenomenological analysis was used to explore, throung semistructured interviews, the lived esxperience of living with OSA and useing CPAP.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Gnocchi, Milan, MI, Italy